CLINICAL TRIAL: NCT06906562
Title: A Phase II Nationwide, Fully Decentralized, Telemedicine Study of Pemigatinib in Adult Patients With Advanced or Metastatic Pancreatic Cancer With FGFR2 Gene Fusions or Other FGFR Genetic Alterations
Brief Title: A Phase II Nationwide, Fully Decentralized, Telemedicine Study of Pemigatinib in Adult Patients With Advanced or Metastatic Pancreatic Cancer With FGFR Genetic Alterations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sameek Roychowdhury (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Sameek Roychowdhury, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23382; NCI-2025-03043 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Advanced Pancreatic Carcinoma; Metastatic Pancreatic Carcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pemigatinib; Magnetic Resonance Spectroscopy; Postmortem Imaging; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pemigatinib Treament (Experimental): Patients receive pemigatinib PO QD on days 1-14 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, CT and/or MRI, and OCT throughout the study. Patients may also undergo whole body bone scans and dilated fundoscopy as clinically indicated.
  Interventions: Drug: Pemigatinib; Procedure: Computed Tomography (CT); Procedure: Magnetic Resonance Imaging; Procedure: Optical Coherence Tomography; Procedure: Bone Scan; Procedure: Ophthalmoscopy

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib will be taken orally with a targeted starting does of 13.5 mg
  Other Names: INCB054828
Procedure: Computed Tomography (CT) — Undergo CT scan
  Other Names: CT scan; CAT Scan; computerized tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI; nuclear magnetic resonance imaging; NMRI; Magnetic Resonance Tomography; MRT
Procedure: Optical Coherence Tomography — Undergo OCT
  Other Names: OCT
Procedure: Bone Scan — Undergo whole body bone scan
  Other Names: Bone Scintigraphy
Procedure: Ophthalmoscopy — Undergo dilated ophthalmoscopy
  Other Names: FS; Fundoscopy

SUMMARY:
This phase II study evaluates how well pemigatinib works for the treatment of adult patients with pancreatic cancer that has spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or has spread from where it first started to other places in the body (metastatic) and that have abnormal changes (alterations) in the fibroblast growth factor receptor (FGFR) gene. FGFR genes are genes that, when altered, can lead to and promote the growth of cancer in patients. Researchers want to test if using pemigatinib can block the function of these abnormal FGFR genes and prevent the tumor from growing and whether treatment can help improve overall quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of single agent pemigatinib in patients with advanced or metastatic pancreas cancer of any histologic classification with FGFR2 gene fusions/translocations.

II. To understand response rate and potential for pemigatinib to benefit patients who have other FGFR alterations including point mutations, extracellular small indels and kinase domain duplications in pancreas cancer.

SECONDARY OBJECTIVES:

I. To further evaluate the efficacy of single agent pemigatinib in each above cohort separately.

II. To characterize the safety and tolerability of single agent pemigatinib.

EXPLORATORY OBJECTIVE:

I. To evaluate dynamics of cell-free deoxyribonucleic acid (DNA) (cfDNA) optimized for monitoring response to pemigatinib and detecting emerging resistance mutations to pemigatinib.

OUTLINE: Patients receive pemigatinib orally (PO) once daily (QD) on days 1-14 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, computed tomography (CT) and/or magnetic resonance imaging (MRI), and optical coherence tomography (OCT) throughout the study. Patients may also undergo whole body bone scans and dilated fundoscopy as clinically indicated. After completion of study treatment, patients are followed up at 30 days, then every 4 months for one year.

ELIGIBILITY:
Inclusion Criteria

Patients with histologically or cytologically confirmed advanced or metastatic pancreatic cancer of any histologic classification at the time of diagnosis

* Written documentation of local or central Clinical Laboratory Improvement Act (CLIA)-certified laboratory determination of FGFR gene fusions/translocations or activating mutations
* The study is open to pancreatic cancer in the following cohorts:

  * Cohort 1: Pancreatic cancer of any histology with FGFR2 fusion/translocation (n, up to 30) who have progressed on or are intolerant to at least one standard of care (SOC) therapy. Prior therapy with a different FGFR inhibitor is not permitted. Patients with concurrent Kirsten rat sarcoma (KRAS) mutations are excluded from this cohort
  * Cohort 2: Pancreatic cancer of any histology with activating point mutations, fusion/translocation (FGFR1,3,4) extracellular small indels, or kinase domain duplications (n, up to 10). Patients must have progressed on or are intolerant to at least one SOC therapy. Prior therapy with a different FGFR inhibitor is not permitted. Patients with concurrent KRAS mutations are permitted in this cohort
* Evidence of measurable or evaluable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Patients must have received at least one prior SOC regimen for advanced/metastatic pancreas cancer. Patients should have had evidence of progressive disease following their prior regimen, or if prior treatment was discontinued due to toxicity must have continued evidence of measurable or evaluable disease. Patients who have received prior treatment with an alternate FGFR inhibitor are not eligible for the study
* Patients with symptomatic central nervous system (CNS) metastases are excluded (because it is unclear how much CNS penetration the drug has). However, asymptomatic patients with history of successfully treated CNS metastases with surgery or radiation and follow up imaging showing stability, can be eligible
* Patients ≥ 18 years of age of either gender
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 (patients with ECOG performance status of 2 may be considered on a case-by-case basis after discussion with Incyte)
* Able to read and/or understand the details of the study and provide written evidence of informed consent as approved by Institutional Review Board (IRB)/Ethics Committee (EC)
* Recovery from adverse events of previous systemic anti-cancer therapies to baseline or Grade 1, except for:

  * Alopecia
  * Stable neuropathy of ≤ Grade 2 due to prior cancer therapy
* Able to swallow and retain oral medication
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests

Exclusion Criteria

* Neurological symptoms related to underlying disease requiring increasing doses of corticosteroids.

  * Note: Steroid use for management of CNS tumors is allowed but must be at a stable dose for at least 2 weeks preceding study entry
* History of another primary malignancy except adequately treated in situ carcinoma of the cervix or non-melanoma carcinoma of the skin or any other curatively treated malignancy that is not expected to require treatment for recurrence during the course of the study or affect survival
* Any other medical condition that would, in the investigator's , prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures
* Current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjuctivitis, confirmed by ophthalmologic examination
* History and/or current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium, and lung with the exception of calcified lymph nodes, minor pulmonary parenchymal calcifications, and asymptomatic coronary calcification
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral pemigatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
* Current evidence of endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis etc.
* Treatment with any of the following anti-cancer therapies prior to the first dose of pemigatinib within the stated timeframes:

  * Cyclical chemotherapy (intravenous) within a period of time that is shorter than the cycle length used for that treatment (e.g., 6 weeks for nitrosourea, mitomycin-C)
  * Biological therapy (e.g., antibodies - including bevacizumab) within a period of time that is ≤ 5 t1/2 or ≤ 4 weeks, whichever is shorter, prior to starting study drug
  * Continuous or intermittent small molecule therapeutics within a period of time that is ≤ 5 t1/2 or ≤ 4 weeks (whichever is shorter) prior to starting study drug
  * Any other investigational agents within a period of time that is ≤ 5 t1/2 or less than the cycle length used for that treatment or ≤ 4 weeks (whichever is shortest) prior to starting study drug
  * Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug
* Patients who are currently receiving treatment with agents that are known strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration are excluded. Patients are not permitted to receive enzyme-inducing anti-epileptic drugs
* Consumption of grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, Seville oranges or products within 7 days prior to first dose
* Absolute neutrophil count (ANC) ≤ 1,000/mm^3 [1.0 x 10^9/L]
* Platelets ≤ 75,000/mm^3 [75 x 10^9/L] • Hemoglobin ≤ 9.0 g/dL
* Total bilirubin ≥ 1.5x upper limit of normal (ULN) unless associated with patient's primary cancer and/or metastases and with principal investigator's approval
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 3x ULN unless associated with patient's primary cancer and/or metastases and with principal investigator's approval
* Alkaline phosphatase ≥ 2.5x ULN unless associated with patient's primary cancer and/or metastases and with principal investigator's approval
* Calculated or measured creatinine clearance of < 40 mL/min
* Calcium-phosphate homeostasis:

  * Inorganic phosphorus outside of institutional normal limits
  * Total serum calcium (can be corrected) outside of institutional normal limits
* History of clinically significant or uncontrolled cardiac disease including unstable angina, acute myocardial infarction, New York Heart Association Class III or IV congestive heart failure, or arrhythmia requiring therapy. Subjects with a pacemaker and well-controlled rhythm for at least 1 month prior to first dose will be allowed
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months following the discontinuation of study treatment. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine systems (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential
* Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after the last dose of the study drug and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via seminal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 24 months
  The proportion of patients with a best overall response of complete response (CR) or partial response (PR). Overall response rate assessed per RECIST v1.1. Will be evaluated in all patients who received at least 80% of the recommended dose of pemigatinib averaged over a 9-week period. ORR will be calculated along with its 95% confidence interval

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 12 months
  PFS will be evaluated in all patients who received at least 80% of the recommended dose of pemigatinib averaged over a 9-week period. Will be analyzed using the Kaplan-Meier method.
Disease Control Rate (DCR) | Up to 12 months
  Defined as the proportion of patients with a best overall response of CR or PR or SD. Will be assessed using descriptive stats. The estimated ORR and corresponding 95% confidence intervals based on the binomial distribution will be reported.
Overall Survival (OS) | Up to 12 months
  OS will be evaluated in all patients who received at least 80% of the recommended dose of pemigatinib averaged over a 9-week period. Will be analyzed using the Kaplan-Meier method.
Type, frequency and severity of adverse events | Up to 12 months
  The severity of AEs will be assessed according to the NCI CTCAE v5.0
Best overall response (BOR) | Baseline up to 1 year after completion of study treatment.
  BOR will be summarized for each cohorts using the ORR and the Disease Control Rate which are the proportion of patients having respectively a best overall response of partial response (PR) or complete response (CR), or stable disease (SD), PR or CR. The estimated ORR and corresponding 95% confidence intervals based on the binomial distribution will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sameek Roychowdhury, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (71):
- United States (71):
  - Ohio State University-Telemedicine, Birmingham, Alabama
  - Ohio State University-Telemedicine, Mobile, Alabama
  - Ohio State University-Telemedicine, Anchorage, Alaska
  - Ohio State University-Telemedicine, Phoenix, Arizona
  - Ohio State University-Telemedicine, Tucson, Arizona
  - Ohio State University-Telemedicine, Hot Springs, Arkansas
  - Ohio State University-Telemedicine, Los Angeles, California
  - Ohio State University-Telemedicine, San Diego, California
  - Ohio State University-Telemedicine, San Francisco, California
  - Ohio State University-Telemedicine, Auroa, Colorado
  - Ohio State University-Telemedicine, New Haven, Connecticut
  - Ohio State University-Telemedicine, Wilmington, Delaware
  - Ohio State University-Telemedicine, Washington D.C., District of Columbia
  - Ohio State University-Telemedicine, Jacksonville, Florida
  - Ohio State University-Telemedicine, Miami, Florida
  - Ohio State University-Telemedicine, Orlando, Florida
  - Ohio State University-Telemedicine, Tampa Bay, Florida
  - Ohio State University-Telemedicine, Atlanta, Georgia
  - Ohio State University-Telemedicine, Augusta, Georgia
  - Ohio State University-Telemedicine, Honolulu, Hawaii
  - Ohio State University-Telemedicine, Boise, Idaho
  - Ohio State University-Telemedicine, Champaign, Illinois
  - Ohio State University-Telemedicine, Chicago, Illinois
  - Ohio State University-Telemedicine, Fort Wayne, Indiana
  - Ohio State University-Telemedicine, Indianapolis, Indiana
  - Ohio State University-Telemedicine, Des Moines, Iowa
  - Ohio State University-Telemedicine, Iowa City, Iowa
  - Ohio State University-Telemedicine, Kansas City, Kansas
  - Ohio State University-Telemedicine, Wichita, Kansas
  - Ohio State University-Telemedicine, Lexington, Kentucky
  - Ohio State University-Telemedicine, New Orleans, Louisiana
  - Ohio State University-Telemedicine, Bar Harbor, Maine
  - Ohio State University-Telemedicine, Baltimore, Maryland
  - Ohio State University-Telemedicine, Boston, Massachusetts
  - Ohio State University-Telemedicine, Ann Arbor, Michigan
  - Ohio State University-Telemedicine, Detroit, Michigan
  - Ohio State University-Telemedicine, Minneapolis, Minnesota
  - Ohio State University-Telemedicine, St Louis, Missouri
  - Ohio State University-Telemedicine, Bozeman, Montana
  - Ohio State University-Telemedicine, Omaha, Nebraska
  - Ohio State University-Telemedicine, Las Vegas, Nevada
  - Ohio State University-Telemedicine, Concord, New Hampshire
  - Ohio State University-Telemedicine, Albuquerque, New Mexico
  - Ohio State University-Telemedicine, Albany, New York
  - Ohio State University-Telemedicine, New York, New York
  - Ohio State University-Telemedicine, Syracuse, New York
  - Ohio State University-Telemedicine, Charlotte, North Carolina
  - Ohio State University-Telemedicine, Raleigh, North Carolina
  - Ohio State University-Telemedicine, Bismarck, North Dakota
  - Ohio State University-Telemedicine, Fargo, North Dakota
  - Ohio State University-Telemedicine, Cincinnati, Ohio
  - Ohio State University-Telemedicine, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Ohio State University-Telemedicine, Oklahoma City, Oklahoma
  - Ohio State University-Telemedicine, Portland, Oregon
  - Ohio State University-Telemedicine, Philadelphia, Pennsylvania
  - Ohio State University-Telemedicine, Pittsburgh, Pennsylvania
  - Ohio State University-Telemedicine, Charleston, South Carolina
  - Ohio State University-Telemedicine, Memphis, Tennessee
  - Ohio State University-Telemedicine, Nashville, Tennessee
  - Ohio State University-Telemedicine, Austin, Texas
  - Ohio State University-Telemedicine, Dallas, Texas
  - Ohio State University-Telemedicine, Houston, Texas
  - Ohio State University-Telemedicine, San Antonio, Texas
  - Ohio State University-Telemedicine, Salt Lake City, Utah
  - Ohio State University-Telemedicine, Burlington, Vermont
  - Ohio State University-Telemedicine, Norfolk, Virginia
  - Ohio State University-Telemedicine, Richmond, Virginia
  - Ohio State University-Telemedicine, Seattle, Washington
  - Ohio State University-Telemedicine, Morgantown, West Virginia
  - Ohio State University-Telemedicine, Milwaukee, Wisconsin

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu